CLINICAL TRIAL: NCT05751811
Title: Effect of Virtual Reality and Music Therapy on Pain Relief in Outpatient Hysteroscopic Operations: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality and Music Therapy on Pain Relief in OPH Operations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Tsz Yan, Yanny, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2022.617
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Pain
Keywords: Pain relief; Hysteroscopy
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality group (Experimental): Participants under Virtual reality group will wear a virtual reality headset with immersive video content during the whole hysteroscopy.
  Interventions: Device: Virtual reality
- Music therapy group (Experimental): Participants under Music therapy group will wear a headphone playing music during the whole hysteroscopy.
  Interventions: Procedure: Music therapy
- Control group (No Intervention): Participants under Control group will proceed with hysteroscopy as usual practise.

INTERVENTIONS:
Device: Virtual reality — The immersive video simulated a magical journey through a calming starry sky on a flying carpet. The headset will play the immersive video content throughout the hysteroscopic procedure; and will stop playing the content as the procedure comes to an end. Participant can adjust the volume of the sound according to her comfort.
  The duration of hysteroscopic operation will be 5 to 20 minutes.
  Arms: Virtual reality group
Procedure: Music therapy — Relaxing and light music will play throughout the hysteroscopic procedure; and will stop playing as the procedure comes to an end. Participant can adjust the volume of the sound according to her comfort.
  The duration of hysteroscopic operation will be 5 to 20 minutes.
  Arms: Music therapy group

SUMMARY:
Outpatient hysteroscopy can serve as a diagnostic procedure to evaluate for abnormal uterine bleeding, such as menorrhagia or postmenopausal bleeding. This study focuses on the therapeutic aspect of outpatient hysteroscopy, such as myomectomy, polypectomy, intrauterine adhesiolysis and removal of lost intrauterine devices, etc. Apart from the conventional polyp scissors and biopsy forceps, there are also emerging hysterscopic tissue removal systems, such as Truclear®, that can decrease the operation time and increase success of outpatient hysteroscopic operations.

On such occasions, the outpatient hysteroscopic operation needs to be re-arranged in an inpatient setting in the operation theatre under regional or general anesthesia. Therefore, improvement in pain management can reduce participants' health care experience, participants' anaesthetic and procedural risks, decrease healthcare costs, and reduce inconvenience to participants.

This randomized controlled trial aims at evaluating the effectiveness of non-pharmacological interventions (virtual reality and music therapy) in pain management during hysteroscopic operations. It can hopefully provide more local clinical data to explore the role of nonpharmacological techniques in pain control, hence improve our participants' experience in hysteroscopic operations and the potential of providing more hysteroscopic operations as an outpatient setting.

DETAILED DESCRIPTION:
Outpatient hysteroscopy can serve as a diagnostic procedure to evaluate for abnormal uterine bleeding, such as menorrhagia or postmenopausal bleeding. This study focuses on the therapeutic aspect of outpatient hysteroscopy, such as myomectomy, polypectomy, intrauterine adhesiolysis and removal of lost intrauterine devices, etc. Apart from the conventional polyp scissors and biopsy forceps, there are also emerging hysterscopic tissue removal systems, such as Truclear®, that can decrease the operation time and increase success of outpatient hysteroscopic operations. However, there are still chances of failure; and the most common reason for procedure failure is pain. The frequently reported causes of pain include manipulation of the cervix with the tenaculum, uterine distension, application of hysteroscopic instruments, and performance of hysteroscopic operations such as hysteroscopic polypectomy. Some factors further enhance the degree of pain experienced, such as nulliparity, post-menopausal status6, cervical stenosis and high anxiety level.

On such occasions, the outpatient hysteroscopic operation needs to be re-arranged in an inpatient setting in the operation theatre under regional or general anesthesia. Therefore, improvement in pain management can reduce participants' health care experience, participants' anaesthetic and procedural risks, decrease healthcare costs, and reduce inconvenience to participants.

The major pain relief modalities include pharmacological and non-pharmacological techniques. The common analgesic agents used are non-steroid anti-inflammatory drugs (NSAID) and opioids; use of which is limited by their contraindications and side effects, such as deranged renal function and nausea. Non-pharmacological options are therefore a safer alternative. Some studies show that music and virtual reality are effective pain control for out-patient hysteroscopy. However, the evidence has been conflicting so far. To date, there was only one published randomized controlled trial regarding the effectiveness of virtual reality in pain management. The study was conducted overseas and limited by small sample size.

This randomized controlled trial aims at evaluating the effectiveness of non-pharmacological interventions (virtual reality and music therapy) in pain management during hysteroscopic operations. It can hopefully provide more local clinical data to explore the role of nonpharmacological techniques in pain control, hence improve our participants' experience in hysteroscopic operations and the potential of providing more hysteroscopic operations as an outpatient setting.

Objective:

The aim of this randomized controlled trial is to evaluate the effectiveness of nonpharmacological interventions (virtual reality or music therapy) in pain management.

Study protocol:

Participants who meet the inclusion criteria will be introduced to the study by a female research assistant on the day of consultation. For those who agreed to join, their demographic data, obstetric and gynecological histories will be obtained using standardized datasheets. During the consultation, consent for the hysteroscopic operations will be obtained according to the current practice by the attending gynaecologist. Written consent of those who are willing to join the study will also be obtained at the same time.

Their past gynaecological history will be obtained. Participants will be randomly assigned using sealed envelopes to 3 groups: (1) Virtual Reality group, or (2) Music group, or (3) Control group (current standard practice with no pain relief during the outpatient hysteroscopic operations). Randomization will be carried out by using block randomization method with 1:1:1 ratio in block size of 6 and stratified by menopausal status (premenopausal or post-menopausal). Due to the nature of the intervention, both the investigators and the participants are not blinded to the allocation.

Participants assigned to the Virtual Reality group will be given the virtual reality headset with immersive video content for use during the whole hysteroscopy. Participants in the music group will be given a headphone playing light music during the whole hysteroscopy. Both groups of participants can adjust the sound volume on their own according to her comfort. We will also make sure that the participant is able to listen to medical staffs' instructions at the sound volume of her choice. Participants are allowed to stop the video or music by removing the headset or headphone at her own will any time or in the event of side effects. On the other hand, participants in the control group will proceed with whole hysteroscopy as usual.

The attending gynaecologist will then perform the diagnostic hysteroscopy, followed by hysteroscopic operations according to the standard procedures. Generally, a 30-degree hysteroscopy with normal saline as distending medium will be inserted through the cervical os into the uterine cavity under direct vision. No cervical dilation is required unless the hysteroscope failed to pass through the cervical os. After passing through the cervical os and entering the uterine cavity, the uterine cavity will be explored systematically. The diagnostic procedure usually lasts for less than 5 minutes. Attending gynaecologist will proceed with hysteroscopic operations according to clinical needs, e.g. endometrial polypectomy for endometrial polyps, IUCD removal, adhesiolysis of intrauterine adhesion, etc. The indicated surgical procedure will not be affected by this trial.

Whether to proceed with hysteroscopic procedure depends on the assessment of the operative feasibility by the attending gynaecologist, e.g. size of lesion, participant's tolerability, etc. If the procedure is deemed not feasible, participant will be arranged a hysteroscopic surgery under regional or general anesthesia in main operation theatre. The usual practice of management of these participants will not be affected by this trial.

Participants will be asked by the attending nurse or investigator to rate their pain score from 0 to 10 at different time-points during diagnostic hysteroscopy and hysteroscopic operations, with a score of 0 indicating pain-free, while a score of 10 indicating worst pain.

The duration of the whole hysteroscopy is defined as from the time of insertion of hysteroscope into the cervical os until the withdrawal of the hysteroscope, which will be recorded. The highest intra-uterine distension pressure with normal saline will also be recorded.

After the hysteroscopy, the attending gynaecologist will be asked to fill out a datasheet recording the details of the hysteroscopic operations done, the subjective difficulty of the procedure, and to what extent virtual reality or music helps with pain relief of the participant on a scale of 0 to 10.

On the other hand, participants will be asked if they have experienced any side effects during the procedure. Besides, participants will be asked to rate their satisfaction towards the mode of pain relief method (if any), the outpatient hysteroscopy in general, the communication with the attending gynaecologist and staff during the hysteroscopy and their acceptance towards outpatient hysteroscopy in the future if indicated. Finally, they will be asked to rate the pain score 30 minutes after their procedure. Follow-up appointment or further treatment will be given to participant, if indicated, and not affected by this trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants scheduled for outpatient hysteroscopy in Prince of Wales Hospital.
* Participants who are willing to give written consent to participate in the study.

Exclusion Criteria:

* Participants who have hearing or visual deficits.
* Participants who cannot understand written Chinese.
* Participants refuse to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of the pain score of virtual reality therapy compared to control group (no intervention) in outpatient hysteroscopy. | up to 1.5 years
  The change of the pain score of virtual reality therapy at different time-point during outpatient hysteroscopy, compared to control group (no intervention).
  Pain score from 0 to 10, with 0 being no pain and 10 the most severe pain.
The change of the pain score of music therapy compared to control group (no intervention) in outpatient hysteroscopy. | up to 1.5 years
  The change of the pain score of music therapy at different time-point during outpatient hysteroscopy, compared to control group (no intervention). Pain score from 0 to 10, with 0 being no pain and 10 the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Yan Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong